CLINICAL TRIAL: NCT06271499
Title: The Effect of Using Smart Glasses Integrated Ultrasonography on the Success of the Procedure and Comfort of the Anesthesiologist in Radial Artery Catheterization
Brief Title: The Effect of Using Smart Glasses Integrated Ultrasonography on Radial Artery Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Collaborators: Ayşegül Güven (Unknown); Bengi Safak (Unknown); Ahmet Onat Bermede (Unknown)
Responsible Party: Principal Investigator, Merve Gozen, Specialist, M.D., Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AnkaraU-Smart-cannulation
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Catheterization; Cannulation
Keywords: Radial artery cannulation; Ultrasonography; Smart glasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Patients underwent radial artery catheterization using standard USG
  Interventions: Other: Radial artery catheterization with USG
- Group II (Active Comparator): Patients underwent radial artery catheterization using smart glasses integrated UGG
  Interventions: Other: Radial artery catheterization with smart glasses integrated UGG

INTERVENTIONS:
Other: Radial artery catheterization with USG — Radial artery catheterization with USG The catheterization was performed by two anesthesiologist with different experience (Junior practitoner who has the experience of 20-50, and the senior practitioner who has the experience of >50 radial artery catheterizations). The side to be catheterized was determined by modifie Allen test which was first performed on the nondominant hand. After general anesthesia induction, a 45° angle was given to wirst of selected side with a support. After skin asepsis, radial artery was vizualized 2 centimeter (cm) above the wrist in short axis with the high-frequency linear USG probe. The radial artery puncture was performed while step by step monitoring the needle tip in short axis out-of-plane technique. Following the puncture, radial artery catheterized with a 3 French 8 cm catheter.
  Arms: Group I
Other: Radial artery catheterization with smart glasses integrated UGG — The catheterization was performed by two anesthesiologist with different experience (Junior practitoner who has the experience of 20-50, and the senior practitioner who has the experience of >50 radial artery catheterizations). Before the study, as practitioners had no previous experience with smart glasses, they performed 5 catheterizations with smart glasses integrated USG on model. The side to be catheterized was determined by modifie Allen test which was first performed on the nondominant hand. After general anesthesia induction, a 45° angle was given to wirst of selected side with a support. After skin asepsis, radial artery was vizualized 2 centimeter (cm) above the wrist in short axis with smart glasses integrated high-frequency linear USG probe. The radial artery puncture was performed while step by step monitoring the needle tip in short axis out-of-plane technique. Following the puncture, radial artery catheterized with a 3 French 8 cm catheter.
  Arms: Group II

SUMMARY:
The use of Ultrasonography (USG) in arterial catheterization, in which the comfort of the practitioner and hand-eye coordination become very important, is frequently needed by anesthesiologists in their daily practice. The aim of this study is to evaluate the success rate and anesthesiologist's satisfaction between two practitioners with different levels of experience in radial artery catheterization with smart glasses USG.

DETAILED DESCRIPTION:
The arterial catheterizations were usually performed by anesthesiologists in operation rooms and intensive care units for many reasons such as blood pressure monitoring and gas sampling. The choice of radial artery is because of its anatomic advantages. However some patients related features can cause difficulties in catheterization. The use of ultrasounography (USG) guidance raises the rate of success and decreases the complications. Coordination skills between hand, eye, procedure area and screen are essential for the USG-guided catheterization. Smarth glasses, project the USG image in real-time directly in front of the practitioner's eyes and thus allows the practitioner to simultaneously view the screen and the procedure area. The primer aim of this study is to evaluate the success rate and anesthesiologist's satisfaction between two practitioners with different levels of experience in radial artery catheterization with smart glasses USG. The secondary aims are to evaluate the cannulation time and complications between groups.

120 patients >18 years who would be undergone elective elective surgery with an indication for radial artery catheterization between August 2022 and December 2022 were included to the prospective, randomised, single centre study. Patients underwent radial artery catheterization for any reason in the last one month, and with contraindications for catheterization were excluded. Patients were divided randomly into two groups (Group I: patients underwent radial artery catheterization using standart USG, and Group II: patients underwent radial artery catheterization using smart glasses integrated UGG). The catheterization was performed by two anesthetists with different experience. The subcutaneous distance, radial artery depth and diameter in short axis, cannulation time and ergonomic satisfaction of the practitioners were recorded. The program SPSS 11.5 was used to analyze data.

ELIGIBILITY:
Inclusion Criteria:

* >18 years who would have undergone elective elective surgery with an indication for radial artery catheterization between August 2022 and December 2022

Exclusion Criteria:

* Patients who underwent radial artery catheterization for any reason in the last 1 month and with contraindications for catheterization

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
The success rate | At the end of the radial artery catheterization
  After the catheterization, when the artery waveform was on monitor, the catheterization was considered successful.
The anesthesiologist's satisfaction | At the end of the radial artery catheterization
  The ergonomic satisfaction of the practitioner was evaluated on a 5-point Likert scale (1: Very dissatisfied, 2: Dissatisfied, 3: Undecided, 4: Satisfied, 5: Very satisfied).

SECONDARY OUTCOMES:
The cannulation time | At the end of the radial artery catheterization
  The time between puncture and the seen of artery waveform seen was recorded as cannulation time
Complications | At the end of the radial artery catheterization
  After catheterization, the radial artery was re-imaged with USG in terms of complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Medical Faculty, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No